CLINICAL TRIAL: NCT03733418
Title: Vitamin D to Improve Outcomes by Leveraging Early Treatment: Long-term Brain Outcomes in Vitamin D Deficient Patients (VIOLET-BUD)
Brief Title: Vitamin D to Improve Outcomes by Leveraging Early Treatment: Long-term Brain Outcomes in Vitamin D Deficient Patients
Acronym: VIOLET-BUD
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); University of Colorado, Denver (Other); Montefiore Medical Center (Other); Intermountain Medical Center (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jin H. Han, Associate Professor, Vanderbilt University Medical Center
Other Study IDs: 181553
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-08

CONDITIONS: Cognitive Decline
Keywords: vitamin D; cognitive decline; dementia; critical care
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Cholecalciferol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention: Patients who received high dose D3 and completed the neuropsychological evaluations at 12 (+/-4) months after randomization.
  Interventions: Drug: 540,000 IU vitamin D3
- Placebo: Patients who received placebo and completed the neuropsychological evaluations at 12 (+/-4) months after randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 540,000 IU vitamin D3 — This intervention was administered as part of VIOLET parent study. A single dose of 540,000 IU vitamin D3 was administered within 2 hours of randomization time.
  Other Names: Cholecalciferol
  Groups: Intervention
Drug: Placebo — Placebo that matched the vitamin D3 color was provided.
  Groups: Placebo

SUMMARY:
This ancillary study will determine if early administration of a single high-dose (540,000 IU) oral vitamin D3 (cholecalciferol) treatment improves 12-month global cognition and executive function as determined by comprehensive neuropsychological testing in 140 critically ill patients with Vitamin D deficiency at enrollment.

DETAILED DESCRIPTION:
VIOLET-BUD is an ancillary study to a parent double-blinded, placebo-controlled randomized control trial (RCT) evaluating how a single, high-dose (540,000 IU) oral Vitamin D3 treatment affects 90-day mortality in patients who are at high risk for ARDS and have Vitamin D deficiency (plasma 25-hydroxyvitamin D < 20 ng/ml) at enrollment. The parent RCT (Vitamin D to Improve Outcomes by Leveraging Early Treatment [VIOLET], NCT03096314) is part of the Clinical Trials Network for the Prevention and Early Treatment of Acute Lung Injury (PETAL) sponsored by the NHLBI. The VIOLET trial completed enrollment in July 2018 with 1,360 randomized to either high dose, enteral Vitamin D3 or placebo.

This ancillary study will provide additional funding to perform comprehensive neuropsychological (cognitive) evaluations, which were not part of the parent trial. These neuropsychological evaluations will be conducted 12 (+/- 4) months after randomization among a subset of 140 survivors enrolled in VIOLET. This ancillary study will conducted in 7 (out of 42) sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled in the VIOLET parent study

Exclusion Criteria:

* Deaf or blind
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 584 patients enrolled in VIOLET.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin H. Han, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (7):
- United States (7):
  - University of Colorado Hospital, Aurora, Colorado
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Montefiore Medical Center, New York, New York
  - Oregon Health and Science University Hospital, Portland, Oregon
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Intermountain Medical Center, Murray, Utah

IPD SHARING:
Plan to Share IPD: Yes
This data sharing plan is only pertinent to data collected specifically for VIOLET-BUD. Because VIOLET-BUD is an ancillary study to a Prevention and Early Treatment of Acute Lung Injury (PETAL) network study, the same data sharing plan will be instituted as the PETAL Clinical Coordinating Center. Limited access data sets will be prepared and provided to the NHLBI in accordance with National, Heart, Lung and Blood Institute (NHLBI) policies on data sharing: http://www.nhlbi.nih.gov/research/funding/human-subjects/set-preparation-guidelines.
  VIOLET-BUD data will be made available on the Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC). In addition to the data, documentation such as data collection forms, study procedures and protocols, data dictionaries and algorithms for calculated data elements and descriptions of all variable recoding performed will also be provided.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available after the publication of the primary manuscript.

REFERENCES:
- [Derived] Han JH, Ginde AA, Brown SM, Baughman A, Collar EM, Ely EW, Gong MN, Hope AA, Hou PC, Hough CL, Iwashyna TJ, Jackson JC, Khan A, Orun OM, Patel MB, Raman R, Rice TW, Ringwood N, Semler MW, Shapiro NI, Talmor DS, Self WH; Vitamin D to Improve Outcomes by Leveraging Early Treatment Network Investigators. Effect of Early High-Dose Vitamin D3 Repletion on Cognitive Outcomes in Critically Ill Adults. Chest. 2021 Sep;160(3):909-918. doi: 10.1016/j.chest.2021.03.046. Epub 2021 Apr 2. PMID 33819472
- See also: Pubmed link to manuscript — https://pubmed.ncbi.nlm.nih.gov/33819472/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D3: Participants randomized to the vitamin D3 group received a single enteral (oral or enteral tube) dose of 540,000 IU vitamin D3 (cholecalciferol).
- Placebo: Patients randomized to the control group received a placebo solution matched in appearance to the vitamin D3 solution.
Period: Overall Study
Arm/Group | Vitamin D3 | Placebo
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 | Placebo | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [39.5 to 65] | 46.0 [37.5 to 63.5] | 53 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 25 | 46
  Male | 26 | 23 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 40 | 31 | 71
  Race: Black or African American | 4 | 8 | 12
  Race: Asian | 1 | 1 | 2
  Race: American Indian or Alaskan Native | 1 | 1 | 2
  Race: Native Hawaiian or other Pacific Islander | 1 | 1 | 2
  Race: Other | 0 | 5 | 5
  Race: Multiple race | 0 | 1 | 1
Facility residence before hospitalization [Count of Participants; unit: Participants]
  Home (independently) | 39 | 39 | 78
  Home (with help) | 5 | 7 | 12
  Home (with professional help) | 2 | 0 | 2
  Nursing facility | 1 | 2 | 3
Dementia [Count of Participants; unit: Participants] | 4 | 4 | 8
Education, y [Median (Inter-Quartile Range); unit: years] | 14 [12 to 16] | 14 [12 to 16] | 14 [12 to 16]
Charlson Comorbidity Index [Median (Inter-Quartile Range); unit: units on a scale] — The Charlson comorbidy index provides takes into account 19 comorbid conditions and assigns a weight for each comorbid condition. It ranges from 0 to 37 points with higher scores representing higher comorbidity burden.
  units on a scale | 3 [1 to 4.5] | 2 [0 to 3.75] | 2 [1 to 4]
Barona Index [Median (Inter-Quartile Range); unit: units on a scale] — The Barona Index estimates intelligence using age, sex, region of residence, years of education, and highest occupation. A score of 100 indicates normal intelligence. A score < 100 indicates below normal intelligence and a score > 100 indicates above normal intilligence.
  units on a scale | 107.7 [101.9 to 112.9] | 109.0 [101.8 to 113.0] | 108.4 [101.7 to 113.1]
SOFA Score [Median (Inter-Quartile Range); unit: units on a scale] — The SOFA score characterizes severity of illness based on the performance of several organ systems in the body: neurologic, blood, liver, kidney, and blood pressure/hemodynamics/vasopressor use. Scores range from 0 to 22 with higher scores representing higher severities of illness.
  units on a scale | 4 [2 to 7] | 5 [2 to 7] | 5 [2 to 7]
Infection (Sepsis + Pneumonia) [Count of Participants; unit: Participants] | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: 12-month Cognition as Measured by the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
Description: The RBANS is a comprehensive neuropsychological battery for the evaluation of global cognition and has been validated in subjects with mild cognitive impairment, moderate to severe traumatic brain injuries, vascular dementias, and Alzheimer's disease. It specifically tests for for immediate and delayed memory, attention, visuospatial construction, and language. Scores range from 0 to 160 with 100 representing the population average. Higher score represents better cognition.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
units on a scale | 79.6 [73 to 84] | 82.1 [74.7 to 84.6]

2. Primary Outcome: 12-month Executive Function as Measured by the Components of the Delis-Kaplan Executive Function System (D-KEFS) Subscales.
Description: The D-KEF's Proverbs, Number-Letter Switching, and Verbal Fluency Category Switching subscales will measure conceptual flexibility, inhibition, and monitoring, respecitvely, which encompasses the majority of executive function. The average of the three subscales will provide an executive function composite score. Scores range from 1 to 18; 10 is considered normal, and higher values indicate better executive function.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
units on a scale | 8.1 [6.8 to 9.0] | 8.7 [7.4 to 9.3]

3. Secondary Outcome: 12-month Functional Status as Measured by Katz Activities of Daily Living (ADL) Scale.
Description: The Katz ADL quantifies basic ADLs such as bathing, dressing, toileting, transferring, continence, and feeding. Scores range from 0 (completely dependent) to 6 (completely independent).
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 6.0 [6.0 to 6.0] | 6.0 [6.0 to 6.0]

4. Secondary Outcome: 12-month Loss of Employment
Description: Loss of employmentwas used using the Outcomes After Critical Illness and Surgery (OACIS) Employment Survey and characterizes the patient's baseline and current (12-month) employment status. Patients were defined as having a loss of employment if they went from full to partial or no employment or partial to no employment at 12 months.
Time Frame: 12 (+/- 4) months
Population: Patients who were partially or fully employed prior to randomization.
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 20 | 29
Participants | 7 | 10

5. Secondary Outcome: All-cause Mortality
Description: Patients were contacted and consented at the same time as the 12-month outcome assessments. Therefore, no patients who were enrolled in VIOLET-BUD died.
Time Frame: 12 (+/- 4) months
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
Participants | 0 | 0

6. Secondary Outcome: Nursing Home Residence at 12-months
Description: Patient resides in a nursing home.
Time Frame: 12 (+/- 4) months
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
Participants | 1 | 1

7. Secondary Outcome: 12-month Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Immediate Memory Domain
Description: Immediate memory is 1 of the 5 cognitive domains tested in the RBANS. Scores range from 40 to 160, with higher scores representing better immediate memory. A score of 100 represents the population average. The standard deviation for the population is 15.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 84.1 [80.2 to 89.0] | 87.6 [83.0 to 93.9]

8. Secondary Outcome: 12-month Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Visuospatial Construction Domain
Description: Visuospatial construction is 1 of the 5 cognitive domains tested in the RBANS. Scores range from 40 to 160, with higher scores representing better visuospatial construction. A score of 100 represents the population average. The standard deviation for the population is 15.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 70.7 [66.0 to 75.9] | 68.7 [64.6 to 73.9]

9. Secondary Outcome: 12-month (Repeatable Battery for the Assessment of Neuropsychological Status) RBANS Language Domain
Description: Language is 1 of the 5 cognitive domains tested in the RBANS.Scores range from 40 to 160, with higher scores representing better language. A score of 100 represents the population average. The standard deviation for the population is 15.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 95.7 [90.1 to 97.4] | 95.6 [90.0 to 97.5]

10. Secondary Outcome: 12-month Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) Attention Domain
Description: Attention is 1 of the 5 cognitive domains tested in the RBANS. Scores range from 40 to 160, with higher scores representing better attention. A score of 100 represents the population average. The standard deviation for the population is 15.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 87.9 [80.7 to 95.0] | 90.1 [82.4 to 96.1]

11. Secondary Outcome: 12-month Delayed Memory Domain
Description: Delayed memory is 1 of the 5 cognitive domains tested in the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS). Scores range from 40 to 160, with higher scores representing better delayed memory. A score of 100 represents the population average. The standard deviation for the population is 15.
Time Frame: 12 (+/- 4) months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 85.1 [81.4 to 91.3] | 84.6 [81.4 to 91.0]

12. Secondary Outcome: Functional Status as Measured by the Lawton Instrumental Activities of Daily Living Scale.
Description: The Lawton IADL quantifies instrumental ADLs such using the telephone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and finances. This scale ranges from 0 (completely dependent) to 8 (completely independent).
Time Frame: 12 months (+/- 4 months)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Vitamin D3 | Placebo
Number analyzed (Participants) | 47 | 48
score on a scale | 8.0 [7.9 to 8.0] | 8.0 [8.0 to 8.0]

ADVERSE EVENTS:
Time Frame: The median follow-up times were 443 days (IQR, 384-484 days) and 442 days (IQR, 401-477 days) in the vitamin D3 and placebo groups, respectively.
Arm/Group | Vitamin D3 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 0/47 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT03733418/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT03733418/SAP_001.pdf